CLINICAL TRIAL: NCT00981526
Title: Telmisartan as an Adjunctive Treatment for Metabolic Problems in Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Xiaoduo Fan, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-P-000790
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Cognition; Metabolism; Antipsychotics; Psychopathology
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Telmisartan; Clozapine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Telmisartan (Experimental): (existing Clozapine or Olanzapine treatment) + (Telmisartan)
  Interventions: Drug: Telmisartan; Drug: Clozapine; Drug: Olanzapine
- B: Placebo (Placebo Comparator): (existing Clozapine or Olanzapine treatment) + (Placebo)
  Interventions: Drug: Placebo; Drug: Clozapine; Drug: Olanzapine

INTERVENTIONS:
Drug: Telmisartan — Telmisartan 40mg/day for the first 2 weeks.
  Telmisartan 80mg/day for the next 10 weeks.
  Arms: A: Telmisartan
Drug: Placebo — Placebo (plus existing clozapine or olanzapine treatment) for 12 weeks.
  Arms: B: Placebo
Drug: Clozapine — Clozapine (plus telmisartan or placebo) for 12 weeks.
Drug: Olanzapine — Olanzapine (plus telmisartan or placebo) for 12 weeks.

SUMMARY:
This is a 12-week, randomized, double-blinded, placebo-controlled trial of telmisartan 80 mg/day as an adjunctive to clozapine or olanzapine therapy, in 70 schizophrenia subjects to examine telmisartan's effect on glucose metabolism, weight, food intake, resting energy expenditure, and body composition. In addition, the study will examine insulin's effects on psychopathology and cognition.

Potential subjects will be identified by their clinicians at the Freedom Trail Clinic, or Massachusetts General Hospital. Approximately 70 subjects will be enrolled.

DETAILED DESCRIPTION:
The specific aims include:

Primary Aims:

1. Examine the efficacy of telmisartan added to regular doses of clozapine or olanzapine in improving insulin resistance.
2. Examine the efficacy of telmisartan in reducing fasting triglycerides.

Secondary Aims:

1. Examine the effects of telmisartan on negative symptoms, positive symptoms, and cognitive function.
2. Examine telmisartan's effects on lipids, body composition, and waist/hip ratio.
3. Examine telmisartan's effects on inflammatory biomarkers including C-reactive protein (CRP) and interleukin 6 (IL-6).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Diagnosis of schizophrenia, any subtype or schizoaffective disorder, any subtype
3. Treatment with clozapine or olanzapine for at least 6 months
4. Stable dose of antipsychotic agent for at least one month
5. Well establish compliance with out-patient medications
6. Females subjects will be eligible to participate in the study if they are of non-childbearing potential or of child-bearing potential and willing to practice appropriate birth control methods (complete abstinence from sexual intercourse, female sterilization, sterilization of male partner, implants of levonorgestrel, injectable progestogen, oral contraceptives, intrauterine devices, or double barrier methods of contraception using spermicide with either a condom or diaphragm) during the study.

Exclusion Criteria:

1. Inability to provide informed consent
2. Current substance abuse
3. Psychiatrically unstable
4. Significant medical illness including severe cardiovascular, hepatic, renal disease
5. Current insulin treatment of diabetes
6. History of immunosuppression
7. Current or recent radiation or chemotherapy treatment for cancer
8. Chronic use of steroids
9. Pregnancy or breast feeding
10. Use of diuretics, digoxin, warfarin because the possible drug-drug interaction of telmisartan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoduo Fan, MD, MPH, MS, Principal Investigator — UMass Medical School
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Fan X, Copeland P, Nawras S, Harrington A, Freudenreich O, Goff DC, Henderson DC. Adjunctive telmisartan treatment on body metabolism in clozapine or olanzapine treated patients with schizophrenia: a randomized, double blind, placebo controlled trial. Psychopharmacology (Berl). 2019 Jun;236(6):1949-1957. doi: 10.1007/s00213-019-5181-z. Epub 2019 Feb 12. PMID 30747254
- [Derived] Fan X, Song X, Zhao M, Jarskog LF, Natarajan R, Shukair N, Freudenreich O, Henderson DC, Goff DC. The effect of adjunctive telmisartan treatment on psychopathology and cognition in patients with schizophrenia. Acta Psychiatr Scand. 2017 Nov;136(5):465-472. doi: 10.1111/acps.12799. Epub 2017 Aug 29. PMID 28851055

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 66 subjects were screened, 4 of which were screen fails. 62 subjects were then enrolled. Prior to randomization, 8 subjects withdrew consent. 54 subjects were randomized.
Groups:
- A: Telmisartan: Telmisartan 80mg/day
- B: Placebo: Placebo
Period: Overall Study
Arm/Group | A: Telmisartan | B: Placebo
Started | 26 | 28
Completed | 22 | 22
Not Completed | 4 | 6
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- B: Placebo: Placebo Group
- Total: Total of all reporting groups
Arm/Group | A: Telmisartan | B: Placebo | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 28 | 54
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.65 (12.14) | 44.68 (11.02) | 43.22 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 23 | 27
  Male | 22 | 5 | 27

OUTCOME MEASURES:

1. Primary Outcome: Insulin Resistance
Description: Insulin resistance as estimated by homeostasis model of assessment of insulin resistance (HOMA-IR) at week 12 in both the experimental and placebo arm. Insulin resistance is a condition in which cells fail to respond to the normal action of the hormone in the body. The HOMA-IR is calculated using a subject's fasting plasma insulin and glucose levels. The higher the score, the higher the level of insulin resistance.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: HOMA-IR scores
Arm/Group | A: Telmisartan | B: Placebo
Number analyzed (Participants) | 22 | 22
HOMA-IR scores | 1.9997 (1.4262) | 2.5824 (2.469)

2. Primary Outcome: Triglycerides
Description: Fasting triglycerides assessed in both experimental and placebo arm at week 12.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | A: Telmisartan | B: Placebo
Number analyzed (Participants) | 22 | 22
mg/dl | 154.15 (156.02) | 176.72 (96.65)

3. Secondary Outcome: Lipid Metabolism - LDL-cholesterol and HDL-cholesterol
Description: Lipid metabolism - fasting low density lipoprotein (LDL) and high density lipoprotein (HDL) are estimated in both experimental and placebo arms at 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- A: Experimental: Telmisartan 80mg/day
Arm/Group | A: Experimental | B: Placebo
Number analyzed (Participants) | 22 | 22
mg/dl
  LDL-cholesterol | 107 (35.71) | 107.85 (31.57)
  HDL-cholesterol | 41.05 (9.59) | 43.18 (11.71)

4. Secondary Outcome: Psychopathology - PANSS Total, PANSS - Negative Score, PANNS - Positive Score and SANS - Total Scores.
Description: The Positive and Negative Syndrome Scale (PANSS) and Scale for the Assessment of Negative Symptoms (SANS) were used to assess the positive and negative symptoms in experimental and placebo arms at 12 weeks. The PANSS total scale includes positive and negative subscales. For both subscales, the score ranges from 7-49 and total PANSS score ranges from 30-210. The total scale is a summation of all the subscales. The SANS score ranges from 0-100. For all scales, a greater score represents a worse outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A: Experimental | B: Placebo
Number analyzed (Participants) | 22 | 22
units on a scale
  PANSS total score | 67.41 (13.36) | 71.05 (20.32)
  PANSS negative score | 19.55 (5.80) | 19.95 (5.09)
  PANSS positive score | 15.50 (5.55) | 16.68 (7.64)
  SANS total score | 27.82 (11.27) | 29.28 (10.96)

5. Secondary Outcome: Body Composition: Waist to Hip Ratio
Description: Body composition as estimated by waist to hip ratio in both experimental and placebo arms at 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | A: Telmisartan | B: Placebo
Number analyzed (Participants) | 22 | 22
Ratio | 0.99 (0.08) | 0.95 (0.23)

6. Secondary Outcome: Body Composition: Percent Total Body Fat
Description: Body composition estimated by percent total body fat as measured by a dual energy absorptiometry (DXA) scan in both experimental and placebo arms at 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | A: Telmisartan | B: Placebo
Number analyzed (Participants) | 22 | 22
percentage of body fat | 31.9 (9.88) | 31.28 (9.02)

ADVERSE EVENTS:
Arm/Group | A: Experimental | B: Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 8/22 | 2/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Experimental (N=22) | B: Placebo (N=22)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dizziness (General disorders) | 3 (3) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No